CLINICAL TRIAL: NCT06224257
Title: A Phase 2, Multicenter, Single-arm, Open-label Study on the Efficacy and Safety of PI3K Inhibitors in Relapsed/Refractory Large Granular T Lymphocytic Leukemia
Brief Title: Efficacy and Safety of Linperlisib in Relapsed/Refractory Large Granular T Lymphocytic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: YL-Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023083
Record Dates: First submitted 2024-01-08; First posted 2024-01-25 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-01

CONDITIONS: Relapsed/Refractory Large Granular T Lymphocytic Leukemia
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Linperlisib (Experimental): Linperlisib was administered at 80 mg every day, orally in a 28-day cycle until disease progression or intolerable toxicity occurred.
  Interventions: Drug: Linperlisib

INTERVENTIONS:
Drug: Linperlisib — Elevated PI3K activity in T-LGL likely plays an important role in the ability of the pathologic cells to avoid homeostatic apoptosis, since inhibition of this pathway leads to apoptosis in the population of cells harboring the pathologic clone. More importantly, the activity of this pathway may represent a kind of "Achilles heel" for T-LGL in that PI3K inhibitors alone are quite effective at inducing spontaneous apoptosis in the clonal CTLs after a short incubation.
  Other Names: PI3K Inhibitor

SUMMARY:
This is a prospective, multicenter, single-arm, phase 2 study. This study aims to evaluate the efficacy and safety of Linperlisib, the PI3K delta inhibitor for patients with relapsed/refractory large granular T lymphocytic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 18 years
* Diagnosis of T-cell large granular lymphocytic leukemia (T-LGLL)
* Meet any of the following indications for treatment： 1. Hemoglobin < 100g/L or RBC transfusion dependence 2. Neutrophil count <0.5×10^9/L or neutrophil count decreased with recurrent infection 3. Progressive splenomegaly and/or Massive Splenomegaly 4. Combined with autoimmune diseases requiring treatment, such as rheumatoid arthritis, autoimmune thyroiditis, etc. 5. Severe B symptoms
* Failure or intolerance to a first-line therapy
* ECOG performance status ≤2
* Expected survival ≥ 6 months
* Willing and able to comply with the requirements for this study and written informed consent

Exclusion Criteria:

* History of other lymphoproliferative neoplasms
* Had malignant tumor within 5 years before enrollment, exclusive of cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial tumor, cervical carcinoma in situ or other indolent tumors
* Previously received organ or stem cell transplantation
* Patients with active infection within 2 weeks before giving the first dose of medication
* Patients with HBV, HCV, HIV or other infections that require treatment
* History of immunodeficiency, or congenital immunodeficiency disorders
* Any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study, including clinically significant cardiac diseases, refractory hypertension, metabolic disorders and other diseases that seriously affect the function of the gastrointestinal tract.
* Abnormal liver function: two consecutive examinations with an interval of ≥1 week suggest that ALT and AST are 2.5 times higher than the upper limit of normal values
* Renal impairment: creatinine clearance <30ml/min
* History of mental illness
* History of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severe impairment of lung function, etc.
* Received attenuated vaccine 4 in weeks before enrollment
* Participation in another clinical trial within 4 weeks before the start of this trial
* Have an allergy to Linperlisib or any other part of this medicine.
* Pregnant or breast-feeding patients
* Patients considered to be ineligible for the study by the investigator for reasons other than the above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2023-12-03 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with hematologic remission | 8-12 weeks
  Hematological response is evaluated by hemoglobin (Hb), absolute neutrophil count (ANC), platelet count (PLT), absolute lymphocyte count (ALC), absolute large granular lymphocyte count, and blood transfusion.

SECONDARY OUTCOMES:
Incidence of the adverse event | 8-12 weeks
  Use Common Terminology Criteria for Adverse Events (CTCAE) Version 5 to assess the adverse event Use Common Terminology Criteria for Adverse Events (CTCAE) Version 5 to assess the adverse event Use Common Terminology Criteria for Adverse Events (CTCAE) Version 5 to assess the adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Jun Shi, PhD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (3):
- China (3):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Zhoukou Central Hospital, Zhoukou, Henan
  - Regenerative Medicine Center, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No